CLINICAL TRIAL: NCT05795452
Title: Environmental Mixtures, Cognitive Control and Reward Processes, and Risk for Psychiatric Problems in Adolescence
Status: Suspended | Type: Observational
Why Stopped: The PI and study are transferring to another institution
Sponsor: Columbia University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAU9473; 5R01ES032296-03 (NIH); 8191 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Psychiatric Problem
Keywords: Functional magnetic resonance imaging (fMRI); Cognitive function; Cognitive Control; Reward Processing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents from the Mothers and Newborns Cohort

SUMMARY:
This study aims to examine the cognitive and neural pathways underlying the joint impact of chemical and social exposures on two aspects of cognitive function: cognitive control and reward processing. The investigators will use high resolution, multi-band resting state and task functional magnetic resonance imaging (fMRI) as well as neuromelanin stain MRI to identify pathways through which exposure to a mixture of prenatal chemical and early life social exposures alters brain function and behavior. Specifically, the investigators will leverage extant prenatal exposure data (N=550) from the Columbia Center for Children's Environmental Health (CCCEH) Mothers and Newborns (MN) birth cohort and study symptoms and brain function in adolescence.

DETAILED DESCRIPTION:
Adolescence is a period of high risk for the emergence of psychiatric issues, particularly attention problems, substance abuse, and psychotic experiences. Risk for these problems likely originates in the prenatal period when the brain undergoes significant rapid change, making this a particularly vulnerable time for alterations in brain development. Few studies have examined risk from prenatal exposure to neurotoxicants that emerge in adolescence and the biological pathways that underlie these associations. Emerging findings suggest that prenatal exposure to environmental chemicals (e.g. environmental tobacco smoke (ETS), air pollutants such as polycyclic aromatic hydrocarbons (PAH)) is associated with behavioral symptoms of attentiondeficit/ hyperactivity disorder (ADHD), substance use disorders (SUD), and psychotic disorders (PD). These symptoms often emerge across adolescence, and frequently co-occur, suggesting shared underlying causes in the brain. Prenatal chemical exposures often co-occur with each other and with social exposures, such as early life stress (ELS) that are also associated with elevated behavioral symptoms. The joint contributions of these chemical and social exposures to these behavioral symptoms are understudied, as are the cognitive and neural pathways linking exposure to behavior.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 13-20 years
* Available prenatal exposure data
* Adolescents and parents are English- or Spanish-speaking

Exclusion Criteria:

* Presence of metallic device or dental braces
* Full Scale Intelligence Quotient (IQ) < 70 at prior assessment
* Pregnant women or lactating women

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The current proposed study is funded to conduct resting state and task fMRI and assessment of psychiatric symptoms in 250 adolescents in the Mothers and Newborns birth cohort. Prenatal exposure data will be leveraged from the CCCEH database.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Youth Self Report (YSR) from the Child Behavior Checklist (CBCL) | 15 minutes during study visit
  This is a 112-question scale for adolescents about their own behavioral functioning. It has a Likert-like scoring format and multiple syndrome and DSM-oriented scales, with higher scores indicating more symptoms. Raw scores are converted to T scores with a mean of 50 and standard deviation of 10. The range is 0 to 90.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Margolis, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - New York State Psychiatric Institute, New York, New York